CLINICAL TRIAL: NCT03929445
Title: A Comparative Study Between Air-Q Intubating Laryngeal Mask And Fastrach Intubating Laryngeal Mask By Using Bougie Assisted Endotracheal Intubation
Brief Title: Bougie Assisted Endotracheal Intubation in Air-Q Intubating Laryngeal Mask And Fastrach Intubating Laryngeal Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Ghada A.Kamhawy, Clinical professor, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ghada
Record Dates: First submitted 2018-11-08; First posted 2019-04-26 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-03

CONDITIONS: Intubation;Difficult; Endotracheal Tube Wrongly Placed During Anesthetic Procedure
Keywords: Bougie; Air Q; Fastrach

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- AIR-Q group (Active Comparator): the group which selected randomly to try AIR-Q device
  Interventions: Device: Endotracheal tube introducers
- I-LMA group (Active Comparator): the group which selected randomly to try I-LMA device
  Interventions: Device: Endotracheal tube introducers

INTERVENTIONS:
Device: Endotracheal tube introducers — Endotracheal tube introducers (gum elastic bougie) for emergency intubation The endotracheal tube introducer (ETI) is an effective and inexpensive adjunct to difficult airway management that is easy to use.
  ETI is solid introducer 60-70 cm long with a 35 - 40 distally angulated (Coude) tip. They are easy to use, widely available, and have been used as adjuncts to difficult direct laryngoscopy for many decades.
  The gum elastic bougie is usually guided by tactile clicks as the device passes the cartilage rings of the trachea. After Supraglottic devices are removed, an ETT can subsequently be railroaded over the bougie.
  Other Names: The Gum Elastic Bougie

SUMMARY:
This study aims to compare using bougie as an assistant for endotracheal intubation through Air-Q and Fastrach intubating laryngeal mask devices when blind intubation fails as attempt to increase its success rate.

DETAILED DESCRIPTION:
The investigators hypothesis that using bougie with its smaller caliber or lesser size can facilitate intubation and improve success rate when blind intubation through both devices fails.

Study objectives

* To make a comparison between Air-Q intubating laryngeal mask and Fastrach intubating laryngeal mask by using bougie assisted endotracheal intubation through both devices in patients undergoing elective surgeries in Suez Canal Hospitals.
* To assess the first trial success rate, the total success rate, time to tracheal intubation, the number of attempts, hemodynamics and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged >18 years old.
* Gender both male and female.
* Patients are ASA I (American Society of Anesthesiologists' physical status Grade I) normal healthy patients or ASA II patients with mild systemic disease and no functional limitations

Exclusion Criteria:

* Any disorder of the cardiovascular, pulmonary, hepatic, renal, or gastrointestinal systems known from history or general examination.
* Patients with unstable cervical spine
* Any medical disease that may affect airway as Rheumatoid arthritis.
* Patient refusal to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
success rate of endotracheal intubation on the first, second and third attempts in both devices Air-Q and fastrach | 180 seconds after anethesia induction
  If the blind intubation is failed through Air Q or Fastrack Intubating laryngeal mask the investigator will use gum elastic bougie to facilitate introducing an endotracheal tube estimation of success rate of endotracheal intubation on the first, second and third attempts
The time needed for devices insertion (Air Q and Fastrach Intubating Laryngeal mask) | !80 seconds after anesthesia induction
  1. Air Q and Fastrach Intubating laryngeal mask insertion time in seconds will be measured (device time).
  2. Endotracheal tube (ETT) insertion time will be measured ( ETT time).
  3. Total insertion time will be estimated (Device Time + ETT Time )

SECONDARY OUTCOMES:
Incidence of adverse events | Intraoperative and in the first 48 postoperative hours
  Incidence of adverse events and complications during and after the procedure will be also recorded. Complications, including laryngospasm, bleeding, false passage, and sore throat will be recorded intraoperatively and in the first 48 postoperative hours.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada A. Kamhawy, Lecturer, Principal Investigator — Suez Canal University
Locations (1):
- Ghada A.Kamhawy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided